CLINICAL TRIAL: NCT03218059
Title: Outcome After MTX & Transvaginal Surgery or UAE & Uterine Curettage in Patients With Cesarean Scar Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-CSP Treatment
Record Dates: First submitted 2017-03-12; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-01

CONDITIONS: Cesarean Scar Pregnancy; Menstruation
Keywords: Cesarean Scar Pregnancy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Methotrexate Combined With Transvaginal Surgery — The methods of treatment of CSP
  Other Names: Uterine Artery Embolization Combined With Uterine Curettage

SUMMARY:
Cesarean scar pregnancy (CSP)is one of the more serious complications of pregnancies that occur after a prior cesarean delivery. No clinical guidelines have been issued for the management of CSP. More than 30 treatment methods are reported to be used in managing CSP. However, which management can achieve better clinical effects remains unknown. Therefore, this prospective study is designed to compare the outcome between MTX + transvaginal surgery and UAE + D&C in the treatment of CSP.

ELIGIBILITY:
Inclusion Criteria:

Increased levels of serum β-hCG and ultrasonography findings. The criteria for diagnosis by ultrasonography was the presence of the following: (1) an empty uterine cavity and endocervical canal; (2) detection of the placenta and/or a gestational sac embedded in the hysterectomy scar; (3) the presence of the gestation sac with or without a fetal pole and with or without fetal cardiac activity (depending on the gestational age) in the anterior part of the uterine isthmus; and (4) a thin (1-3 mm) or absent myometrial layer between the gestational sac and the bladder. All patients had taken Magnetic Resonance Imaging (MRI) to clarify the diagnosis . Pregnancy tissues were identified by histopathology examinations of the surgical tissues.

Exclusion Criteria:

All enrolled patients had no contraindications for transvaginal surgery or UAE, including renal failure, active pelvic infection, clotting disorders, or known allergy to the contrast material.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Duration of menstruation by questionnaire | six months after treatment
  Duration of menstruation
Endocrine level by blood examination | six months after treatment
  FSH in IU/L
Volume of menstruation by questionnaire | six months after treatment
  in pictorial blood loss score

SECONDARY OUTCOMES:
The length of the CSD by MRI | six months after treatment
  millimeter
The depth of the CSD by MRI | six months after treatment
  millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, Study Chair — Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University
Locations (1):
- Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University, Shanghai, Shanghai Municipality, China